CLINICAL TRIAL: NCT00276510
Title: Efficacy and Tolerance of EGb 761® 120mg Two Times a Day on Dementia of Alzheimer Type's Onset in Patients Suffering From Memory Complaints. A Randomised, Double-blind, Multicentre, Parallel Groups, Placebo Controlled Phase IIIb/IV Study in Elderly Over 70
Brief Title: A Study of EGb 761® (Tanakan®) in Dementia of Alzheimer Type Onset in Patients Suffering From Memory Complaints
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-31-00240-011
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Memory Disorders, Age-Related; Retention Disorders, Cognitive
MeSH Terms: conditions — Memory Disorders | interventions — Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: EGb 761® (Tanakan®)
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: EGb 761® (Tanakan®) — 120 mg, 1 tablet twice a day, oral route, during 5 years.
  Arms: 1
Other: Placebo — 1 tablet twice a day, oral route, during 5 years.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Tanakan® is effective at slowing the progression from memory complaint to dementia of Alzheimer's type.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneously reporting a memory complaint
* Short anxiety battery test < 6, (only if patient screened at GP site)
* Geriatric depression scale < 15
* Mini-mental state (MMS) > 25 in GP's office (in hospital site MMS is done as complementary scale)

Exclusion Criteria:

* Objective memory impairment
* Clinician rated dementia staging system > 0.5
* Mini-mental state < 25
* Dementia, past history of seizures, Parkinson disease

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2878 (Actual)
Dates: Start 2002-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
EGb 761® efficacy on conversion rate of memory complaint to dementia of Alzheimer type by a survival analysis | Baseline, month 12, 24, 36, 48 and 60

SECONDARY OUTCOMES:
Efficacy on rate of cognitive abilities decline | Baseline, month 12, 24, 36, 48 and 60
Effect on concomitant diseases | Baseline, month 12, 24, 36, 48 and 60
Concomitant treatments' reports | Baseline, month 12, 24, 36, 48 and 60
Global evaluation of memory complaint by the patient | Baseline, month 12, 24, 36, 48 and 60
Clinical safety | Baseline, month 12, 24, 36, 48 and 60

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (696):
- France (696):
  - 1 rue de l'Orient, Agde
  - 3 Avenue de Marlioz, Aix-les-Bains
  - 3 rue Auguste Delaune, Alès
  - 17 rue du Cardinal Georges d'Amboise, Amboise
  - 17 rue Manuel, Amboise
  - 83 rue Nicolas et Paul Paquet, Ancerville
  - 10 bd De La Republique, Andernos-les-Bains
  - 107 bd De La Republique, Andernos-les-Bains
  - 19 rue Jean Saccheti, Andernos-les-Bains
  - 128 Rue Bressigny, Angers
  - 18 rue Martin Luther King, Angers
  - 2 boulevard Jacques Millot, Angers
  - 21 bd Roi René, Angers
  - 25, rue St Nicolas, Angers
  - 59 Boulevard Joseph Bédier, Angers
  - 61 Ave Jean XXIII, Angers
  - 68A rue d'Orgemont, Angers
  - Residence le Paradis Bat 17, 74-78 rue Volney, Angers
  - Centre Hospitalier Universitaire Hotel Dieu Gerontologie Clinique 4 rue Larrey, Angers
  - 111 rue de la Chalouère, Angers
  - 4 rue Saint Jacques, Angers
  - 4, rue St Jacques, Angers
  - 7 rue Thiers, Angers
  - 1172 route de Grasse Ste Elisabeth, Antibes
  - 20 boulevard Albert 1er, Antibes
  - 700 av. Jules Grec, Antibes
  - 26 R Pres Wilson, Ars-sur-Moselle
  - Avenue Joseph Lafont, Aubagne
  - Groupe Piettot Bâtiment 2, Aubagne
  - 37-39 boulevard Anatole France, Aubervilliers
  - 26 av. Charles de Gaulle, Aubevoye
  - 3 Avenue de Verdun, Audenge
  - 27 rue Maréchal Foch, Aumetz
  - 2 bis route de Miremont, Auterive
  - 70 bis rue Etienne Billieres, Auterive
  - 17 rue des Ecoles, Avoine
  - 17, rue des Ecoles, Avoine
  - 10 Allée Des Rochers, Avrillé
  - 30 Ter Avenue Pierre Mendès, Avrillé
  - 5 Place Maréchal Juin, Avrillé
  - Rd point de Gal de Gaulle, Avrillé
  - 1 Résidence Marcel Paul, Bachant
  - 11 rue du pont Fouchard, Bagneux
  - 13, rue Denis Papin, Bagnolet
  - 11 rue du Général Cheroutre, Bailleul
  - 17 rue de la Croix de Pierre, Bain-de-Bretagne
  - 9 av Pierre Coupeau, Balma
  - 43 rue Ducs de Bar, Bar-le-Duc
  - 33 rue Jean Jaures, Bassens
  - 21, rue Georges Clémenceau, Baugé
  - 24, rue Julien Daillière, Bauné
  - Centre Commercial Tertifume 9 rue de Montreuil, Beaucouzé
  - 42 rue de la Petite Porte, Beaufort-en-Vallée
  - 14 rue Moulin du Roy, Beaulieu-sur-Layon
  - L'Helvetia 10 rue Paul Doumer, Beaulieu-sur-Mer
  - 31, rue du Parc, Beaumont-en-Véron
  - Rue Lapeyrère, Beaumont-sur-Lèze
  - 2 r Des Muriers, Beauzelle
  - 24bis, rue de la Motte, Bersée
  - Route de Toulouse, Bérat
  - 1 Avenue Gambetta, Béziers
  - 1, rue du Pinot, Béziers
  - Centre Médical Sémard 39, place Semard, Béziers
  - 9 bis Chemin Aussonne, Blagnac
  - 208 Cours Saint Louis, Bordeaux
  - 28 bd Du President Wilson, Bordeaux
  - 8, Boulevard Albert 1er, Bordeaux
  - Centre Hospitalier Pellegrin-Tripode Service de Neurologie Place Amelie Raba-Leon, Bordeaux
  - Résidence Mozart- Apt 56, 2 rue Jean Artus, Bordeaux
  - 183 Cours De La Marne, Bordeaux
  - Les Suriaux Rue du Stade, Boucé
  - 2 allée Port Larron, Bouchemaine
  - 60 Rue Du Moulin, Bouguenais
  - 1 Rue Roeckel, Bourg-la-Reine
  - 12 Esplanade du Prado, Bourges
  - 121 Avenue du Général de Gaulle, Bourges
  - 14 rue Calvin, Bourges
  - 16 rue Emile Martin, Bourges
  - 24 Boulevard Clémenceau, Bourges
  - 86 Avenue Haegelen, Bourges
  - Centre Hospitalier Jacques Coeur Hopital Taillegrain Centre de Gerontologie des Pres Fichaux 6 rue Taillegrain, Bourges
  - Centre Hospitalier Jacques Coeur Hôpital Taillegrain, Bourges
  - 9, rue du Lavoir, Brain-sur-Allonnes
  - 106, rue du Docteur Lahaye, Breteuil
  - 30 rue de Bayeux, Bretteville-l'Orgueilleuse
  - 1 rue mar Leclerc, Broglie
  - Avenue du Gal de Gaulle, Bruges
  - 57 impasse des Cades, Cabrières
  - 114, rue Authie, Caen
  - 29 rue Lucien Nelle, Caen
  - 36, Avenue Du 6 Juin, Caen
  - 6 Avenue Du 6 Juin 1944, Caen
  - 98 Boulevard du Maréchal Lyautey, Caen
  - Hopital Cote de Nacre Service de Neurologie avenue de la cote de Nacre, Caen
  - Hôpital Côte de Nacre, Caen
  - 12 Grand Rue, Calmont
  - 16, rue d'Alger, Cambrai
  - Square la Gare, Candé
  - Avenue Buchholz, Cantaleu
  - 8 Boulevard Ronceray, Cantenay-Épinard
  - 3 rue Lucien Cassagne, Carbonne
  - La Chohonniere Im. la Rotonde, Carquefou
  - 10 avenue Victor Hugo, Cassis
  - 4 route de Toulouse, Castelmaurou
  - 2 rue Clairval, Castelnau-le-Lez
  - 311 chemin Draye du Marbre, Castelnau-le-Lez
  - Avenue A Briand, Castelnau-le-Lez
  - Villa 54. Résidence le Village, Castelnau-le-Lez
  - Place d'Armes, Cazères
  - 27 rue Emile Landais, Chacé
  - 15 rue des Sables, Chalonnes-sur-Loire
  - 8 rue Seguin, Château Gontier Bazouges
  - 8 rue Sainte Croix, Châteaugiron
  - 16 Bis rue Cherré, Châteauneuf-sur-Sarthe
  - 48 rue Henri Bouriché, Chemellier
  - 290 rue du Bocage, Cheux
  - 11 rue du 11 Novembre 1945, Chinon
  - Place Pierre Robbe, Chinon
  - 14 rue Faidherbe, Cholet
  - 16 Av de l'Europe, Cholet
  - 18, avenue des Calins, Cholet
  - 25 av de Nantes, Cholet
  - 43 Bis Rue Nationale, Cholet
  - 6 Allée des forgerons, Cholet
  - 83 Rue du Paradis, Cholet
  - 55, rue Eugène Lecoq, Clary
  - 7 rue du Docteur Doussain, Clisson
  - 5 rue du Couderc, Colomiers
  - 7 rue d'Auch, Colomiers
  - 13 rue du Docteur Malabouche, Cournonterral
  - 4 Bld Jean-Baptiste Oudry, Créteil
  - 61 Rue de l'amiral Courbet, Croix
  - 9 rue Peyrere, Cubzac-les-Ponts
  - 14 rue du Cezerou, Cugnaux
  - 14, rue Cézerou, Cugnaux
  - 3 avenue de Toulouse, Cugnaux
  - 6 place de Vivier, Cugnaux
  - 2 rue Abbé Bernier, Daon
  - 116 rue Henri Barbusse, Denain
  - 221 rue Villars, Denain
  - 25 place de I'Eglise, Déville-lès-Rouen
  - 11 rue Principale, Diebling
  - 1 Avenue Edouard VII, Dinard
  - 10 rue Mathieu de Dombasle, Dombasle-sur-Meurthe
  - La Tour des Charmettes, Domène
  - 18, rue Danton, Drancy
  - 97, rue Winston Churchill, Dunkirk
  - Résidence Emeraude 71 av Adolphe Geeraert, Dunkirk
  - 72 rue Saint Pierre, Durtal
  - 2 rue Jean Monnet, Eaunes
  - 4 rue du Général de Gaulle, Essey-lès-Nancy
  - Route Nationale 75, Eyguians
  - 108 Faubourg Ambrail, Épinal
  - 3 Place de l'Eglise, Étalondes
  - 1 rue du Jardin Botanique, Évreux
  - 24, rue des Lombards, Évreux
  - 41 rue Victor Hugo, Évreux
  - 6 Centre Commercial les Peupliers, Évreux
  - 7 rue Pasteur, Fabrègues
  - 3 route de Caen, Falaise
  - 33 rue du Camp Fermé, Falaise
  - 2 rue de I'Eglise, Fenouillet
  - 1 rue Renelles, Fécamp
  - 126 Route d'Harcourt, Fleury-sur-Orne
  - 11 bis av. Ambroise Croisat, Fontaine
  - 3 place Louis Maisonnat, Fontaine
  - 1, rue Pierre et Marie Curie, Fontès
  - 21 rue Nationale, Forbach
  - 34 rue du Marechal Soult, Fresnes
  - 2 pl Clemenceau, Fresnes-en-Woëvre
  - 10, Rue Du 8 Mai, Fronton
  - 10 route des Mares, Frossay
  - 74 avenue de la Liberation, Frouard
  - 2 avenue des Camelias, Gan
  - 2 bis rue Abon, Gap
  - 2 bis rue d'Abon, Gap
  - Residence Le Gaughin Bat 1 68 rue Borely, Gardanne
  - Villa Pinede Route St Tropez, Gassin
  - 12 rue Cohue, Gennes
  - 18, avenue de Verdun, Gémenos
  - 24, rue de la République, Gémenos
  - 10 rue de la Sèvre, Gétigné
  - 18 r Stade, Gironde-sur-Dropt
  - 4 ave de la Gare, Gourdan-Polignan
  - Centre Commercial Malartic, Gradignan
  - 41, rue Saint-Yves, Grand-Champ
  - 12, Place Jean Moulin, Grenoble
  - 13 bis rue du General Champon, Grenoble
  - 15, chemin Joseph Brun, Grenoble
  - 22 av. Leon Blum, Grenoble
  - 28 rue Elie Cartan, Grenoble
  - 35 Bd Marechal Foch, Grenoble
  - 46 boulevard Joseph Vallier, Grenoble
  - 6, Boulevard Joseph Vallier, Grenoble
  - 9A place Saint-Bruno, Grenoble
  - Centre de Prevention des Alpes 3 place de Metz, Grenoble
  - 28 rue Général Ferrié, Grenoble
  - 32 rue Gay-Lussac, Grenoble
  - 34 avenue de l'Europe Immeuble le Trident A1er etage, Grenoble
  - 4 avenue de la Bouexiere, Guérande
  - 117 cours de Verdun, Gujan-Mestras
  - 117, avenue du Maréchal de Lattre de Tassigny, Gujan-Mestras
  - 6 pl Du Marché - La Hume, Gujan-Mestras
  - 14 rue de la Liberation, Halluin
  - 14 rue Libération, Halluin
  - 3, rue Paul Vaillant Couturier, Haulchin
  - 12 rue de Maubeuge, Hautmont
  - 206 rue Gambetta, Hautmont
  - 1 rue Franz Schubert Saint Martin d'Hères, Hères
  - 136 av. Ambroise Croizat Saint Martin d'Heres, Hères
  - 20 av. Paul Eluard, Hères
  - 137 Route de Dax, Hinx
  - 2 bis, route de Belin, Hostens
  - 5 rue Mairie, Ingrandes
  - 10 rue Gaston Monmousseau, Ivry-sur-Seine
  - Hopital Charles Foix Service de Gerontologie 37 avenue de la Republique, Ivry-sur-Seine
  - 6 rue des Ponts, Jort
  - 20 avenue de l'Amiral Courbet, Juan-les-Pins
  - 117 Boulevard du Président Wilson, Juan-les-Pins
  - 4 Chemin du Tanit, Juan-les-Pins
  - Le Tanagra- 10 pl du Pont du Lys, Juan-les-Pins
  - 7 Route de Gagnebert, Juigné sur Loire
  - 119 rue Franchepre, Jœuf
  - 2 rue Roger Salengro, L'Haÿ-les-Roses
  - 76, avenue Gabriel Péri, L'Haÿ-les-Roses
  - Le Moulin, La Bâtie-Neuve
  - 33 rue Georges Clemenceau, La Bernerie-en-Retz
  - La buffaie Route du Doreur, La Breille-les-Pins
  - Avenue du Général de Gaulle, La Calmette
  - Maison Médicale av. Géneral de Gaulle, La Calmette
  - 53 rue Martin Luther King, La Chapelle
  - 4 rue Meriadec Laennec, La Chapelle-Basse-Mer
  - 4 rue Mériadec Laënnec, La Chapelle-Basse-Mer
  - 10 rue Aristide Briand, La Chapelle-Heulin
  - 17 rue de l'Erdre, La Chapelle-sur-Erdre
  - 53 rue Martin Luther King, La Chapelle-sur-Erdre
  - 10 , rue Adolphe Abeille, La Ciotat
  - 62, ru du Maréchal de Lattre de Tass, La Forêt-sur-Sèvre
  - 8 Chemin des Vendéens, La Jubaudière
  - 149 route de Bouguenais, La Montagne
  - 9 av. de la Liberation, La Montagne
  - 9 rue de la Liberation, La Montagne
  - Village Retraite, La Motte-du-Caire
  - 4 route de Balaruc, La Peyrade
  - 11 Place Sainte Anne, La Riche
  - 7 route Targon, La Sauve
  - 1 rue Joffre, La Teste-de-Buch
  - 4 place de la République, La Trinité
  - 16 Grand'rue, La Tronche
  - 24 boulevard de la Chantourne, La Tronche
  - 8 Place Vincent Auriol, Labarthe-sur-Lèze
  - 4, chemin Banque, Labastidette
  - 34, rue Vacheresse, Lagny-sur-Marne
  - 23 avenue Pasteur, Laragne-Montéglin
  - 23 rue Louis Pasteur, Laragne-Montéglin
  - 23 rue Pasteur, Laragne
  - 52 Place de la Fontaine, Laragne
  - 43 rue Raymond Poincaré, Laxou
  - 44 bis rue Paul Bert, Laxou
  - 44b rue Paul Bert, Laxou
  - 49 r Theophile Gautier, Le Bouscat
  - 5 Av. Gauthier Lagardère, Le Bouscat
  - 26 Avenue Jean Macé, Le Cailar
  - 8 Avenue Louis Blanc, Le Cailar
  - 6 rue Colbert, Le Canet
  - 1 rue des Orangers, Le Cannet
  - 50 Bd Sadi Carnot, Le Cannet
  - 69 av. F. Roosevelt, Le Cannet
  - Route de Marignac, Le Fousseret
  - 7 place du Commerce, Le Fuilet
  - 17 rue du Dr Leveillé, Le Grand-Pressigny
  - 35 Avenue du Président Kennedy, Le Grand-Quevilly
  - 60 rue des Moussaillons, Le Grau-du-Roi
  - 1 Quai de Bretagne, Le Lion-dAngers
  - 1 rue Pasteur, Le May
  - 48 rue des Mauges, Le Mesnil-en-Vallée
  - 111 route de Paris, Le Mesnil-Esnard
  - Impasse Mérite, Résidence Lamiot rue L'ecalier, Le Neubourg
  - 31 rue Promenade, Le Puy-Saint-Bonnet
  - 21 rue de Nantes, Le Temple-de-Bretagne
  - 364 rue Pasteur, Le Versoud
  - 23 rue Jeanne d'Arc, Les Epesses
  - 46 rue de Paris, Les Lilas
  - 2 rue des Pleiades, Les Mureaux
  - 8 Avenue Amiral Chauvin, Les Ponts-de-Cé
  - 68 ter Rue Marjolin, Levallois-Perret
  - 11 place de l'Eglise, Lherm
  - 34 avenue Georges Clémenceau, Libourne
  - 46 avenue François Mitterand, Liffré
  - 110 BD de la liberté, Lille
  - 115 bis rue d'Artois, Lille
  - 129 Rue Des Postes, Lille
  - 19 Rue Des Postes, Lille
  - 236 rue du Faubourg des Postes, Lille
  - 24 rue P. Legrand, Lille
  - Hopital Roger Salengro Service de Neurologie C rue Emile Laine, Lille
  - Hôpital Roger Salengro, Lille
  - Parc du Segrais, Lognes
  - 928 avenue de Dunkerque, Lomme
  - Place de la Halle, Longages
  - 2, Rue Abbée Rappine, Longeville-lès-Saint-Avold
  - 47, rue Racine, Longué-Jumelles
  - 126 Avenue des Graves, Lormont
  - 126 Avenue des Gravières, Lormont
  - 126 rue des Gravieres, Lormont
  - 36 avenue de Leuze, Loudun
  - 15 ter Bd Clémenceau, Louviers
  - 57 rue Dupont de l'Eure, Louviers
  - Chemin des Diligences, Louvigné-de-Bais
  - 70 rue Andre Auguste, Lunel-Viel
  - L'ancien Presbytere, Lussan-Adeilhac
  - 10, avenue Robert Daugey, Luynes
  - 1 Place Bellecroix, Manduel
  - 1 bis avenue des Coteaux, Marly
  - 2 Avenue Long Pré, Marly
  - 8 Rue Georges Thiebaux, Mars-la-Tour
  - 1 boulevard Montricher, Marseille
  - 134, rue Félix Pyat, Marseille
  - 81 rue Jaubert, Marseille
  - 12 Bld Des Neiges, Marseille
  - 325 avenue de Mazargues, Marseille
  - 38 bld Rodocanachi, Marseille
  - 431 avenue de Marzargues, Marseille
  - 63, boulevard Rabateau, Marseille
  - Hopital St Joseph Service de Neurologie 26 boulevard Louvain, Marseille
  - 2 Avenue Jean Bouin, Marseille
  - 2 chemin de Morgiou, Marseille
  - 23 Bd de la Concorde, Marseille
  - 250 Bd Romain Rolland, Marseille
  - Groupe Medical de Mazargues 1 av de la Martheline, Marseille
  - 13 rue St Eloi, Marseille
  - 90 Boulevard de Saint Loup, Marseille
  - Les Camoins 58 Traverse de St Menet, Marseille
  - 21 Traverse des Rosiers, Marseille
  - 253 ch. de la Madrague-Ville, Marseille
  - Hopital STe Marguerite Unite de Neurologie 270 boulevard de STe Marguerite, Marseille
  - 6 av. des martyrs de la Resistance, Martignas-sur-Jalle
  - 5 Avenue du Pdt Allende, Martigues
  - Espace Vénitien 1 av Pres Salvador Allende, Martigues
  - Espace Vénitien, Martigues
  - 75 rue Principale, Mazé
  - 1 Square Chardin, Meaux
  - Centre Commercial La Verriere place Beauval, Meaux
  - 11 rue des Tilleuls, Mercy-le-Bas
  - Hôpital Felix Marechal 1 rue Xavier Roussel, Metz
  - 203 Rue de Vallieres, Metz
  - 10 rue de la Republique, Meudon
  - 41, Avenue Plaine Fleurie, Meylan
  - 7 rue de l'Oisans, Meylan
  - Domus Médica, Mèze
  - 206 av de l'Argonne, Mérignac
  - 2 bis Place du Castellas, Milhaud
  - 27 rue de la Croix Thomas, Miniac-Morvan
  - 32 rue Cité, Miré
  - 12 Rue Du 8 Mai 1945, Moirans
  - 221 R de Pont A Mousson, Montigny-lès-Metz
  - 5 rue des Roses, Montigny-lès-Metz
  - 2 place de L'Eglise, Montjean-sur-Loire
  - 2, rue Delpech, Montpellier
  - 25 av de St Lazare - Le Prieure II, Montpellier
  - 32 avenue G Clémenceau, Montpellier
  - 32, Avenue Georges Clémenceau, Montpellier
  - 41 Bld Du Jeu de Paume, Montpellier
  - 7 ter rue Rigaud, Montpellier
  - 82 avenue d'Assas, Montpellier
  - 82, avenue d'ASSAS, Montpellier
  - 9 avenue d'Assas, Montpellier
  - 9, Avenue d'Assas, Montpellier
  - 11 rue Monge, Montpellier
  - 11 rue Mongre, Montpellier
  - 20 avenue de Toulouse, Montpellier
  - 48 rue Robespierre, Montpellier
  - 57, route de Lavérune, Montpellier
  - 59 av. de Toulouse- Bat B, Montpellier
  - 7 rue du Grau, Montpellier
  - 12 Faubourg Boutonnet, Montpellier
  - 22 Faubourg Boutonnet, Montpellier
  - Hopital Gui de Chauliac 80 rue Augustin Fliche, Montpellier
  - 8 rue Pierre Mendès France, Montreuil-Juigné
  - 9 rue Sadi Carnot, Montrouge
  - 113 Route de Douai, Mouchin
  - 11 Rue du Maine, Mouliherne
  - 6, route d'Anjou, Mouliherne
  - 18 Rue de Metz, Moulin Les Metz
  - Rue du Rieu, Moussac
  - 13 rue Clémenceau, Moûtiers
  - 48, ave Jacques Douzans, Muret
  - 48, avenue Jacques Douzans, Muret
  - 25 rue Valentin Desormeaux, Mûrs-Erigné
  - 34 Rue de Metz, Nancy
  - 82 rue Saint Georges, Nancy
  - 15 rue Jeanne d'Arc, Nantes
  - 181 rue Paul Bellamy, Nantes
  - 2 Bd Amiral Courbet, Nantes
  - 23 rue Racine, Nantes
  - 29 bis rue Pelleterie, Nantes
  - 46 bis bd Gabriel Guist'Hau, Nantes
  - 59 bld Gaston Serpette, Nantes
  - 71 rue du Coudray, Nantes
  - 88 rue Gambetta, Nantes
  - Hopital Bellier Service de Geronotologie 41 rue Curie, Nantes
  - 42 rue du Roi Baco, Nantes
  - 7 rue Blancho, Nantes
  - Cabinet de Neurologie - Consultations, Nantes
  - 101 bld de Doulon, Nantes
  - 134 rue du Croissant, Nantes
  - 142 bld Robert Schuman, Nantes
  - 15 rue Guillaume Grootaers, Nantes
  - 23 bld Chauviniere, Nantes
  - 27 boulevard des Americians, Nantes
  - 34 rue de la Gourmette, Nantes
  - 46, boulevard Jules Verne, Nantes
  - 58 bld Jules Verne, Nantes
  - 63 rue de la Bottière, Nantes
  - Route de Morlaas, Navailles-Angos
  - 12 rue Pasteur, Neuville-sur-Escaut
  - 12, rue Pasteur, Neuville-sur-Escaut
  - 16 rue Vernier, Nice
  - 30, rue Gioffredo, Nice
  - 54 bld François Grosso, Nice
  - 6, rue Rossini, Nice
  - Hopital de Cimiez Pavillon Mossa 4 avenue de la Reine Victoria, Nice
  - Hôpital Pasteur, Nice
  - 32 rue Auguste Gal, Nice
  - 47 Bis, Rue Barberis, Nice
  - 5 boulevard du General Delfino, Nice
  - 5 rue Smolett, Nice
  - L'Esperanza 9 rue de la République, Nice
  - Maison Médical Mutualiste, Nîmes
  - Centre Raymond Ruffi 12 rue Alexandre Ducros, Nîmes
  - Cabinet Medical place des Goelands, Nîmes
  - 30 Bd de la Gare, Nort-sur-Erdre
  - 4 bld de Strasbourg, Nort-sur-Erdre
  - 8 rue Foch, Novéant-sur-Moselle
  - 20 Place d'Armes, Nueil-les-Aubiers
  - 2 Allée des Glycines, Orly
  - 2 avenue Pesqué, Orthez
  - 2, Avenue Pesqué, Orthez
  - 3 rue Madame, Orthez
  - 125, rue Gambetta, Ouistreham
  - 16 rue Aristide Briand, Pacy-sur-Eure
  - 31 rue Jean L'olive, Pantin
  - route de Gizeux, Parçay-les-Pins
  - 19 boulevard Morland, Paris
  - 1 rue Villersexel, Paris
  - 6 rue de la Motte-Piquet, Paris
  - 88 rue de Sevres, Paris
  - 9 Rue de Montessuy, Paris
  - 3, Rue Pierre Le Grand, Paris
  - 40 rue du Faubourg Montmartre, Paris
  - 15 rue de Chabrol, Paris
  - 41 rue de la Grange aux Belles, Paris
  - 26, rue Picpus, Paris
  - 167, boulevard Vincent Auriol, Paris
  - 74 rue Dunois, Paris
  - Hôpital Broca - Service de Gérontologie Clinique 54-56 rue Pascal, Paris
  - 191 rue d'Alésia, Paris
  - 2 rue de la Briqueterie, Paris
  - 96 avenue Maine, Paris
  - 81, rue de Rome, Paris
  - 33, rue Marx Dormoy, Paris
  - 34 rue Hermel, Paris
  - 13 Villa Curial, Paris
  - 20, rue du Télégraphe, Paris
  - 7 Rue Saint Blaise, Paris
  - 79 rue Boissiere, Paris
  - 1 Avenue Mirabelle, Pau
  - 28 rue Castelnau, Pau
  - 69 rue du 14 Juillet, Pau
  - Centre Hospitalier des Pyrenees Department de Psychogeriatrie 29 av du Marechal Leclerc, Pau
  - Centre Hospitalier des Pyrénées, Pau
  - 153 Avenue du Général Leclerc, Pessac
  - 2, rue de l'Hôtel de Ville, Pérols
  - Le forum, Pignan
  - 1 Impasse Pasteur, Pinsaguel
  - 83 rue Andorre, Pinsaguel
  - 18 place Gambetta, Podensac
  - 14 Rue Philippe de Gueldres, Pont-à-Mousson
  - 170 , avenue des Etats-Unis, Pont-à-Mousson
  - 47, boulevard Ney, Pont-à-Mousson
  - 7 rue du Cardinal Mathieu, Pont-à-Mousson
  - 3 bis rue Cacheleux, Pont-de-l'Arche
  - 35bis rue du Général de Gaulle, Pont-de-l'Arche
  - 26, rue de Tourte, Pornic
  - 1 place Aristide Briand, Pornichet
  - 16 av. du Littoral Ste Marguerite, Pornichet
  - Immeuble "Le Roc Rose", Port-de-Bouc
  - 69 rue du Général Leclerc, Potigny
  - 69, rue du Général Leclerc, Potigny
  - 169 , rue de l'Avenir, Poulx
  - BP 22-23 rue republique, Preignac
  - 24 avenue Charles de Gaulle, Pulnoy
  - 7 rue Gambetta, Quarouble
  - Cours Goudouli, Quint-Fonsegrives
  - 141 rue Roger Salengro, Raimbeaucourt
  - 12, rue Louis Braille, Ramonville-Saint-Agne
  - 22 avenue de Tolosane, Ramonville-Saint-Agne
  - 22 avenue Tolosane, Ramonville-Saint-Agne
  - La Garenne, Rauzan
  - 11, rue du Fresne, Renazé
  - Rue Fresnes, Renazé
  - 15 rue Emile Souvestre, Rennes
  - Cabinet de Neurologie 4 av Charles Tillon, Rennes
  - Cabinet de Neurologie, Rennes
  - Centre Commercial La Bellangerais, Rennes
  - Centre Espace Performance, Rennes
  - 3, Rue de la petite Mairie, Restigné
  - Immeuble Athéna 62 bis rue Aristide Briand, Rezé
  - 11 rue Sagazan, Rieumes
  - 9 Place de la Mairie, Roquemaure
  - Quai le Repos, ZAC St Estève, Roquevaire
  - 13 rue de Messan, Rouans
  - 91 avenue Jean Lebas, Roubaix
  - 106 bis Rampe Bouvreuil, Rouen
  - 45 Boulevard de l'Yser, Rouen
  - Hôpital Charles Nicolle Department de Neurologie 1, rue de Germont, Rouen
  - 102 rue Méridienne, Rouen
  - 6 rue Soye, Sains Orens de Gameville
  - 7 place Cambronne, Saint Sebastein Sur Loire
  - 19, Avenue de Verdun, Saint Serin
  - 59 Pl. Du 11 Novembre 1918, Saint-Amand
  - 61 rue Anatole France, Saint-Amand-Montrond
  - Rue des Oratoires, Saint-Anastaise
  - 30 Avenue du Général de Gaulle, Saint-Avertin
  - 4, rue Manet, Saint-Barthélemy-d'Anjou
  - 245, avenue Mindin, Saint-Brevin-les-Pins
  - 13 rue du Commandant Thoreux, Saint-Briac-sur-Mer
  - 4 rue Orme, Saint-Broladre
  - 103 rue Fleurie, Saint-Cyr-sur-Loire
  - 60, Impasses des deux moulins, Saint-Georges
  - 106, Place du Gué des Joncs, Saint-Georges-de-Montaigu
  - 2 rue du Prieuré, Saint-Georges-des-Groseillers
  - 6, rue de Courpouyran, Saint-Georges-dOrques
  - Rue de Clairdouy, Saint-Georges-dOrques
  - 15 bis Avenue Marcellin Berthelot, Saint-Gilles
  - 30 bis avenue Gallieni, Saint-Girons
  - Boulevard du Général de Gaulle, Saint-Girons
  - 2 impasse Dublin, Saint-Herblain
  - 22 av. des Thebaudieres, Saint-Herblain
  - 27 rue d'Aquitaine, Saint-Herblain
  - ZA la Petite Croix, Saint-Hilaire-de-Chaléons
  - 5 rue Daniel Casanova Le Parc des Amandiers, Saint-Jean-de-Védas
  - 11 Route de La Foret, Saint-Jean-des-Linieres
  - 48 avenue Condamine, Saint-Just
  - 22 avenue du Général Leclerc Les Bougainvillées, Saint-Laurent-du-Var
  - 53 Bd du 8 mai 1945, Saint-Macaire-en-Mauges
  - Impasse Dr Adrien Gory, Saint-Mamert-du-Gard
  - 1 Place du 11 Novembre, Saint-Mandrier-sur-Mer
  - 3, Rue Du 3 Août 1944, Saint-Mars-du-Désert
  - 34 rue Prieuré, Saint-Martin-du-Bois
  - 38 rue Hector Berlioz, Saint-Max
  - 63 rue Alexandre 1er, Saint-Max
  - 9, Résidence Haut Rivage, Rue Jean Xxiii, Saint-Max
  - 69 avenue Montaigne, Saint-Médard
  - 112 av Montesquieu, Saint-Médard-en-Jalles
  - 15, avenue Montaigne, Saint-Médard-en-Jalles
  - 107 rue de Pornichet, Saint-Nazaire
  - 3, rue du Pertuischaud, Saint-Nazaire
  - 9, Route du Fort de l'Eve, Saint-Nazaire
  - 1 bis rue Godillot, Saint-Ouen
  - 4, avenue du Petit Montrevault, Saint-Pierre-Montlimart
  - 50 rue Bosq, Saint-Pierre-sur-Dives
  - 1 rue Canot, Saint-Privat-la-Montagne
  - Avenue du 14 Juillet, Saint-Quentin-la-Poterie
  - 16, Boulevard Darby - Valescure, Saint-Raphaël
  - 2, rue Jean Jaurès, Saint-Sébastien
  - 25, avenue de la Martellière, Saint-Sébastien
  - 1 allee Jean Restout, Saint-Sébastien-de-Morsent
  - Route Lombez, Sainte-Foy-de-Peyrolières
  - 146 av de la République, Sainte-Foy-la-Grande
  - 3 rue Moulin du Pain, Sainte-Gemmes
  - Quart Thermal, Salies-de-Béarn
  - 6 Allee Du Merlot, Saussan
  - 30 rue de la Vallee, Sautron
  - 30 rue Vallée, Sautron
  - 1, Allée du Mistral, Savigny-le-Temple
  - 21 rue Chatonnay, Savonnières
  - Place du Port, Segré
  - 3 place de la Gare, Sens-de-Bretagne
  - 72, route Châtel, Sercœur
  - 2 route de Sauvagnon, Serres Castets
  - 14 rue Boltar, Seysses
  - 60 route d'Ox, Seysses
  - 11 rue Football, Sète
  - 12 rue Gabriel Péri, Sète
  - 41 rue Pierre Sémard, Sète
  - 9 rue Alsace Lorraine, Sète
  - Résidence Tarentelle Place E. Herriot, Sète
  - 12 rue Jean Boyer, Sérifontaine
  - 22 Place du Docteur Robert, Sisteron
  - 41 rue Faidherbe, Somain
  - 43, rue Faidherbe, Somain
  - 10 rue Benoît Malon, Sotteville-lès-Rouen
  - 33 rue Littre, Sotteville-lès-Rouen
  - 63 Chaussée du Sillon, St-Malo
  - 27 rue Gaston Chéreau, Thouars
  - 1 Ave des Erables, Tiercé
  - 1 Chemin Courperron, Tilly-sur-Seulles
  - 1 rue de l'Ecotay, Tinténiac
  - 1 Rue des Deportés, Toufflers
  - 1, rue des Ecoles, Toufflers
  - 60 av Du 8 Mai 1945, Toulenne
  - 11 rue De Metz, Toulouse
  - 2, rue Paradoux, Toulouse
  - 26 av. Jean Rieux, Toulouse
  - 35 rue Remusat, Toulouse
  - 68 allee Jean Jaures, Toulouse
  - 76 allee Jean Jaures, Toulouse
  - Centre Hospitalier de Purpan Service de Neurologie place du Docteur Baylac, Toulouse
  - 135 rue Henri Desbals, Toulouse
  - 3 rue Vincent Van Gogh, Toulouse
  - 3 rue Vincent Van Gough, Toulouse
  - 25 Bld des minimes, Toulouse
  - 3 rue Saint Famille, Toulouse
  - 44 av Etienne Billieres, Toulouse
  - 48 all. Charles de Fitte, Toulouse
  - 52 av. de Grande Bretagne, Toulouse
  - 8 pl. Interieure St Cyprien, Toulouse
  - 1 rue Notre Dame, Toulouse
  - 14 rue Jean Duplessis, Toulouse
  - 2 Boulevard Griffoul Dorval, Toulouse
  - 25 av. Marcel Langer, Toulouse
  - 28 rue des Arts, Toulouse
  - 28, rue des Arts, Toulouse
  - 40, bouleard des Récollets, Toulouse
  - 7 avenue Frizac, Toulouse
  - 12 rue Jean Poncelet, Toulouse
  - 150 avenue Jean Chaubet, Toulouse
  - 23, rue Limayrac, Toulouse
  - 24 av. du Cimetiere, Toulouse
  - 44 av. Leon Blum, Toulouse
  - 53 r Du Faubourg Bonnefoy, Toulouse
  - 7 pl Commerciale Jolimont, Toulouse
  - 7 rue Raymond Boulogne Batiment C- apt 23, Toulouse
  - 1 et 3 rue Maryse Bastié, Tours
  - 1, rue Maryse Bartié, Tours
  - 11 rue de Clocheville, Tours
  - 15 rue Jacques Marie Rouge, Tours
  - 2 rue du Plat d'Etain, Tours
  - 26 rue Boisdenier, Tours
  - 29 Bis rue Roger Salengro, Tours
  - 3 rue Victor Hugo, Tours
  - 31, rue Léon Boyer, Tours
  - 63 rue Léon Boyer, Tours
  - 8 rue de Montbazon, Tours
  - 89 rue Jean-Jacques Noirmant, Tours
  - 110 rue de Jemmapes, Tours
  - 5 rue de la Halle, Treviere
  - 26 rue Victor Hugo, Tullins
  - 14 Place de l'Eglise, Uchaud
  - Avenue Georges Chauvin, Uzès
  - Batiment Le Sirius place des Cordeliers, Uzès
  - Hotel des Cordeliers, Uzès
  - Hôtel les Cordeliers place des Cordeliers, Uzès
  - Maison de retraite publique Centre de Memoire Route de Nimes, Uzès
  - Hotel les Cordeliers place des Cordeliers, Uzès
  - route de Montpellier, Vailhauquès
  - 16 rue Anatole France, Valenciennes
  - Res. Saly-2 rue S. Lebourg, Valenciennes
  - 11, Boulevard de la République, Valras-Plage
  - 23 Bd de l'Europe, Vandœuvre-lès-Nancy
  - 12 Place de la République, Varces
  - Le Mistral II, Vauvert
  - 5 avenue de Libourne, Vayres
  - 12 lotissement Figeac, Venerque
  - 41 rue de la Pomme d'Or, Verneuil-sur-Avre
  - 3 Rue Fontaine, Verny
  - Rue de la Poste, Vers-Pont-du-Gard
  - 18 rue de Noailles, Versailles
  - 57 rue Charles Lecour, Vertou
  - 7 rue Mortaliere, Vertou
  - 4 rue du Chapelet, Vezins
  - 15 rue du Jard, Vicherey
  - 5 rue des Halles, Vieillevigne
  - 200 rue Jean Jaures, Vieux
  - 4 Rue Beaurepaire, Vihiers
  - 145 rue de Chevilly, Villejuif
  - 1 bis avenue Outrebon, Villemomble
  - 8 Av G. Clémenceau, Villenave-d'Ornon
  - 8 Av. du Gal Clémenceau, Villenave-d'Ornon
  - Centre Commercial Chamboparc, Villenave-d'Ornon
  - 164 boulevard des Fontaines, Villeneuve-lès-Maguelone
  - 1 Rue René Cassin, Villeneuve-Tolosane
  - 22, rue du Maréchal Foche, Villerupt
  - 1, rue des Charmes, Villette-d'Anthon
  - 10 Chemin Vignes d'Oule, Villevêque
  - 88 rue Liverdun, Villey-Saint-Étienne
  - Rue du 8 Mai 1945, Vinay
  - 3 avenue Segond, Vincennes
  - 56, avenue de Paris, Vincennes
  - 11 rue du Faton, Voiron
  - 15 route de la Gare, Vourey
  - 9, place Sainte Anne, Vue
  - 85 rue Jean Jaurès, Vue
  - 64 avenue du 14 Juillet, Wattignies
  - Maison Medicale Bichat, Wattrelos

REFERENCES:
- [Derived] Vellas B, Coley N, Ousset PJ, Berrut G, Dartigues JF, Dubois B, Grandjean H, Pasquier F, Piette F, Robert P, Touchon J, Garnier P, Mathiex-Fortunet H, Andrieu S; GuidAge Study Group. Long-term use of standardised Ginkgo biloba extract for the prevention of Alzheimer's disease (GuidAge): a randomised placebo-controlled trial. Lancet Neurol. 2012 Oct;11(10):851-9. doi: 10.1016/S1474-4422(12)70206-5. Epub 2012 Sep 6. PMID 22959217